CLINICAL TRIAL: NCT00003954
Title: Allogeneic Stem Cell Transplantation For Multiple Myeloma: A Two Step Approach To Reduce Toxicity Involving High Dose Melphalan and Autologous Stem Cell Transplant Followed By PBSC Allografting After Low Dose TBI
Brief Title: Melphalan and Stem Cell Transplant Before Total-Body Irradiation and Donor Stem Cell Transplant in Treating Patients With Stage I-III Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1383.00; NCI-2012-00670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA078902 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-04-15 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2019-05

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Bone Marrow Transplantation; Transplantation; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Cyclosporine; Mycophenolic Acid

ARMS (1):
- Treatment (Melphalan and PBSCT before TBI and Donor PBSCT) (Experimental): CONDITIONING REGIMEN: Patients receive high-dose melphalan IV over 15-20 minutes on day -2.
  TRANSPLANTATION: Patients undergo autologous bone marrow or PBSCT on day 0.
  NON-MYELOABLATIVE CONDITIONING REGIMEN: Beginning 40-120 days after autologous transplant, patients undergo TBI on day 0.
  TRANSPLANTATION: Patients undergo donor PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine IV BID on days -1 and 0 and PO BID on days 1-80 with taper based on evaluation of disease response and GVHD. Patients also receive mycophenolate mofetil PO BID on days 0-27.
  POST TRANSPLANT DLI: Beginning 4 weeks after immunosuppression, patients achieving persistent or progressive disease may undergo DLI over 30 minutes every 4 weeks for up to 3 treatments.
  Interventions: Drug: melphalan; Procedure: autologous hematopoietic stem cell transplantation; Procedure: autologous bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation; Drug: cyclosporine; Drug: mycophenolate mofetil; Biological: therapeutic allogeneic lymphocytes

INTERVENTIONS:
Drug: melphalan — Given IV
  Other Names: Alkeran; CB-3025; L-PAM; L-phenylalanine mustard; L-Sarcolysin
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous bone marrow or PBSCT
Procedure: autologous bone marrow transplantation — Undergo autologous bone marrow or PBSCT
  Other Names: ABMT; bone marrow transplantation, autologous; transplantation, autologous bone marrow
Procedure: peripheral blood stem cell transplantation — Undergo autologous bone marrow or PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Procedure: peripheral blood stem cell transplantation — Undergo donor PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Drug: cyclosporine — Given IV and PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Biological: therapeutic allogeneic lymphocytes — Undergo DLI
  Other Names: ALLOLYMPH

SUMMARY:
In this study donor bone marrow transplantation is divided into a two step process to try to significantly reduce the side effects of the procedure yet still provide patients with multiple myeloma the benefits of this procedure

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate engraftment of human leukocyte antigen (HLA) identical peripheral blood stem cell (PBSC) allografts given after conditioning with total-body irradiation (TBI) (200 cGy) and post-grafting immunosuppression with cyclosporine (CSP)/mycophenolate mofetil (MMF) in myeloma patients initially cytoreduced with high-dose melphalan.

II. To evaluate non-relapse mortality at day 100 post allografting. III. To evaluate the efficacy of this allografting strategy in terms of long-term progression free survival (PFS).

OUTLINE:

CONDITIONING REGIMEN: Patients receive high-dose melphalan intravenously (IV) over 15-20 minutes on day -2.

TRANSPLANTATION: Patients undergo autologous bone marrow or PBSC transplantation (PBSCT) on day 0.

NON-MYELOABLATIVE CONDITIONING REGIMEN: Beginning 40-120 days after autologous transplant, patients undergo TBI on day 0.

TRANSPLANTATION: Patients undergo donor PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine IV twice daily (BID) on days -1 and 0 and orally (PO) BID on days 1-80 with taper based on evaluation of disease response and graft-versus-host disease (GVHD). Patients also receive mycophenolate mofetil PO BID on days 0-27.

POST-TRANSPLANTATION DONOR LYMPHOCYTE INFUSION (DLI): Beginning 4 weeks after immunosuppression, patients achieving persistent or progressive disease may undergo DLI over 30 minutes every 4 weeks for up to 3 treatments.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Meet Salmon and Durie criteria for initial diagnosis of multiple myeloma; transplant will be offered to patients with stage II or III multiple myeloma (MM) at diagnosis or have received chemotherapy and/or radiation therapy for progressive MM after initial diagnosis of stage I disease
* The patient must have the capacity to give informed consent
* Have received at least 4 cycles of conventional dose chemotherapy for MM
* DONOR: HLA genotypically identical sibling
* DONOR: Donor must consent to filgrastim (G-CSF) administration and leukapheresis for both peripheral blood stem cell (PBSC) allograft and subsequent DLI
* DONOR: Donor must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral, subclavian)
* DONOR: Age < 75, older donors may be considered after consultation by Psychological Consultation Center (PCC)

Exclusion Criteria:

* Karnofsky score less than 60, unless due solely to myeloma
* Left ventricular ejection fraction less than 40%
* Bilirubin greater than 2 X the upper limit of normal
* Serum glutamic pyruvic transaminase (SGPT) and serum glutamic oxaloacetic transaminase (SGOT) > 2 X the upper limit of normal
* Diffusion lung capacity of carbon monoxide (DLCO) < 50% (corrected) or receiving continuous supplemental oxygen
* Patients with poorly controlled hypertension
* Pregnancy
* Seropositive for the human immunodeficiency virus
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Creatinine clearance < 40 cc/min at the time of initial autografting evaluation
* Prior autograft (can be treated on alternative protocol)
* DONOR: Identical twin
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Infection with human immunodeficiency virus (HIV)
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet Fred Hutchinson Cancer Research Center (FHCRC) criteria for stem cell donation as described in the standard practice guidelines of the institution

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 1999-03; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
PFS | From the date of transplant until the time of progression, relapse, death, or the date the patient was last known to be in remission, up to 3 years
  The current study will be regarded as potentially efficacious if the observed 3-year PFS rate among all patients treated exceeds 30%. The Kaplan-Meier (KM) estimate of PFS will be used.
Decrease in the short-term transplant-related mortality | Day 100 after allograft
Establish stable allogeneic engraftment (mixed or full donor chimerism) | At day 56 after allografting

SECONDARY OUTCOMES:
Overall survival | Up to 3 years
  Estimated by the method of Kaplan and Meier. Confidence intervals will be estimated.
Relapse rate | Up to 3 years
  Summarized using cumulative incidence estimates. Confidence intervals will be estimated.
Response rate | Up to 3 years
  Confidence intervals will be estimated.
Ability to convert mixed to full donor chimerism with DLI | Up to 3 years
  Confidence intervals will be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (4):
- United States (3):
  - City of Hope, Duarte, California
  - University of Colorado, Denver, Colorado
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- University of Torino, Torino, Italy

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241